CLINICAL TRIAL: NCT02016742
Title: A Phase I, Open-label, Randomised, 3-way Crossover Study to Characterise and Compare the Pharmacokinetics, Safety and Tolerability of RDC5 Given as a Single Dose to Healthy Volunteers
Brief Title: A Phase 1 Study of the Pharmacokinetics of RDC5 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chronos Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: RDC5-1-01; 2013-003335-29 (EudraCT Number)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- RDC5 dose level 1 (Experimental): Single dose of RDC5
  Interventions: Drug: RDC5
- RDC5 dose level 2 (Experimental): Single dose of RDC5
  Interventions: Drug: RDC5
- RDC5 dose level 3 (Experimental): Single dose of RDC5
  Interventions: Drug: RDC5
- RDC5 dose level 4 (Experimental): Single dose of RDC5
  Interventions: Drug: RDC5

INTERVENTIONS:
Drug: RDC5

SUMMARY:
The purpose of this study is to characterise the pharmacokinetics, safety and tolerability of RDC5 given as a single dose to healthy volunteers at a number of different dose levels

DETAILED DESCRIPTION:
This is an open-label, randomised, single dose, 3-way crossover study to characterise and compare the PK, safety and tolerability of RDC5 in 15 healthy male volunteers. Eligible subjects will undergo 3 Treatment Periods, each separated by a washout period at least 14 days. Subjects will receive a single dose of RDC5 during each of the three Treatment Periods in line with their randomized treatment sequence. A total of 4 dose levels will be evaluated within the study, though each subject will only receive 3 doses. A Data Review Team (DRT) will review the pharmacokinetic (PK) data from Treatment Periods 1 and 2 and select the doses to be evaluated in Treatment Periods 2 and 3. Subjects will return for a follow visit 21 days after the last dose of RDC5.

ELIGIBILITY:
Inclusion Criteria:

* Willing to use effective method of contraception
* Non smoker or ex-smoker within the previous 6 months

Exclusion Criteria:

* History or presence of any clinically significant findings upon screening
* Participation in a New Chemical Entity clinical study within the previous 124 days or a marketed drug clinical study within the previous 93 days
* Positive result for human immunodeficiency virus (HIV) and/or hepatitis B or C test
* Positive result for urine alcohol and drug screen
* Blood donation ≥ 450 mL in the previous 12 weeks
* Receipt of prescription medicines and/or St John's Wort in the previous 2 weeks

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) for the whole blood concentration of RDC5 | Up to 6 days post dose

SECONDARY OUTCOMES:
AUC from time 0 to time of last observed concentration (AUC0-t) | Up to 6 days post dose
Maximum observed concentration (Cmax) | Up to 6 days post dose
Time at which Cmax occurred (tmax) | Up to 6 days post dose
Elimination half-life (t1/2) | Up to 6 days post dose
Terminal phase elimination rate constant (λz) | Up to 6 days post dose
Apparent volume of distribution (Vd/F) | Up to 6 days post dose
Apparent oral clearance (CL/F) | Up to 6 days post dose
Number (%) healthy volunteers with treatment emergent adverse events (AEs) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, United Kingdom